CLINICAL TRIAL: NCT05712720
Title: A Randomized, Double-Masked, Placebo-Controlled, Parallel-Arm Study to Evaluate the Efficacy and Safety of RZ402 in Participants With Diabetic Macular Edema (DME)
Brief Title: Study to Evaluate the Efficacy and Safety of RZ402 in Diabetic Macular Edema (DME)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Rezolute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: RZ402-201
Record Dates: First submitted 2023-01-17; First posted 2023-02-03 (Actual); Last update posted 2025-10-03 (Actual); Status verified 2025-10

CONDITIONS: Diabetic Macular Edema
Keywords: Diabetic Macular Edema; Diabetic Retinopathy; Diabetes; Retinal; Macular Thickening; Plasma Kallikrein Inhibitor
MeSH Terms: conditions — Diabetic Retinopathy; Diabetes Mellitus

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Group 1 - 50 mg RZ402 (Experimental): RZ402 50mg oral tablet, once daily for 3 months
  Interventions: Drug: Experimental: Group 1 - 50mg RZ402
- Group 2 - 200 mg RZ402 (Experimental): RZ402 200mg oral tablet, once daily for 3 months
  Interventions: Drug: Experimental: Group 2 - 200mg RZ402
- Group 3 - 400 mg RZ402 (Experimental): RZ402 400mg oral tablet, once daily for 3 months
  Interventions: Drug: Experimental: Group 3 - 400mg RZ402
- Group 4 - Placebo (Placebo Comparator): placebo oral tablet, once daily for 3 months
  Interventions: Other: Placebo: Group 4 - Placebo

INTERVENTIONS:
Drug: Experimental: Group 1 - 50mg RZ402 — RZ402 50 mg oral tablet, once daily for 3 months
  Arms: Group 1 - 50 mg RZ402
Drug: Experimental: Group 2 - 200mg RZ402 — RZ402 200mg oral tablet, once daily for 3 months
  Arms: Group 2 - 200 mg RZ402
Drug: Experimental: Group 3 - 400mg RZ402 — RZ402 400mg oral tablet, once daily for 3 months
  Arms: Group 3 - 400 mg RZ402
Other: Placebo: Group 4 - Placebo — Placebo oral tablet, once daily for 3 months
  Arms: Group 4 - Placebo

SUMMARY:
The objective of this trial is to assess the safety, efficacy, and tolerability of RZ402 in patients with Diabetic Macular Edema.

DETAILED DESCRIPTION:
Diabetic macular edema (DME) is a common retinal microvascular complication in diabetic patients that can lead to progressive loss of visual acuity and ultimately to complete vision loss. DME is the main cause of vision loss in patients with Type 2 diabetes. There is a significant unmet medical need to develop better therapies of DME and diabetic retinopathy (DR). RZ402 is a potent and selective plasma kallikrein inhibitor (PKI), which is being developed as an oral therapy for the chronic treatment of DME and DR.

This is a Phase 2, Randomized, Double-Masked, Placebo-Controlled, Parallel-Arm Study to Evaluate the Efficacy and Safety of RZ402 in Participants with Diabetic Macular Edema (DME). A screening period of up to 4 weeks will evaluate eligibility. Once enrolled, patients will be randomized with a 1:1:1:1 ratio to receive RZ402 or placebo for up to 12 weeks. After completing dosing, the patient will enter into a 4 week follow up period.

ELIGIBILITY:
Inclusion Criteria:

General Inclusion Criteria:

1. Confirmed diabetes mellitus Type 1 or Type 2
2. Stable glycemic control

   Study Eye Inclusion Criteria:
3. Mild to moderate non-proliferative diabetic retinopathy (NPDR) with retinal thickening due to CI-DME as determined by the Investigator.
4. Spectral Domain Optical Coherence Tomography (SD-OCT) foveal CST at screening measuring ≥320 µm (or corresponding values)
5. Best Corrected Visual Acuity ETDRS letter score at 4 meters of ≤78 letters at screening.
6. Media clarity, pupillary dilation, and participant cooperation sufficient for adequate clinical evaluations, OCT images and fundus photographs, at screening.

   Fellow Eye Inclusion Criteria:
7. Best Corrected Visual Acuity ETDRS letter score at 4 meters of ≥5 letters at screening.

   Exclusion Criteria:

   Study Eye Exclusion Criteria:
8. Received more than 3 anti-VEGF injections (including Avastin) and/or received a recent anti-VEGF injection within 8 weeks of Randomization.
9. Any history of retinal surgery or other surgical intervention for DME.
10. Intraocular surgery (including cataract surgery), within 12 weeks prior to Randomization, or anticipated need for ocular surgery during the study period.
11. History of trabeculectomy or other filtration surgery (prior laser trabeculoplasty and placement of iStent®1 in conjunction with cataract surgery is permitted if the procedure took place ≥12 weeks prior to Randomization).
12. Autoimmune idiopathic inflammatory eye disease such as anterior uveitis, or participants with history or signs of chronic inflammation.
13. Full thickness macular hole or retinal detachment.
14. Panretinal, macular focal, or grid laser photocoagulation within 16 weeks of Randomization or anticipated need for the use of laser photocoagulation during the study period.
15. Uncontrolled glaucoma, at screening, defined as IOP ≥25 mmHg.
16. The use of corticosteroids as follows:

    1. Topical corticosteroids within 12 weeks prior to Randomization and throughout the remainder of the study.
    2. Use of intraocular or sub-Tenon's steroids within 2 years of Randomization in phakic eyes or 9 months of Randomization in pseudophakic eyes, and throughout the remainder of the study.

    Fellow Eye Exclusion Criteria:
17. Intraocular or sub-Tenon's steroid injection within 6 months of Randomization and throughout the remainder or the study.

    General Exclusion:
18. Use of the following medications or substances within the specified timeframes below and throughout the remainder of the study.

    a. Within 16 weeks of Randomization: i. Systemic anti-VEGF or pro-VEGF treatments ii. Systemic, approved, or off-label drugs or devices used to treat DME iii. Participated in an investigational drug or device study within 16 weeks or 5 half-lives (whichever is longer) of Randomization, including systemic or ocular studies iv. Initiation of drugs or substances known to improve or worsen macular edema e.g., Latanoprost or phosphodiesterase-5 (PDE-5) inhibitors (e.g., Sildenafil or others in PDE-5 class), but participants may remain on these drugs if they were initiated >16 weeks prior to Randomization.

    b. Within 12 weeks of Randomization: i. Use of tobacco- or nicotine- containing products (e.g., cigarettes, cigars, chewing tobacco, snuff, vaping).

    c. Within 4 weeks of Randomization: i. Anti-coagulants, except for aspirin ≤325 mg/day and/or clopidogrel ≤75 mg/day (or equivalent drug class) ii. Total daily doses of Metformin >1000 mg iii. Total daily doses of niacin (Vitamin B3) >1.5 g/day iv. Use of systemic steroids at supraphysiologic doses (e.g., prednisone equivalent of 5 mg/day or hydrocortisone equivalent of 20 mg/day).

    v. Drugs that may affect the retina or optic nerve such as quinolones, thioridazine, deferoxamine, ethambutol, vigabatrin, and pentosan.
19. Alanine aminotransferase (ALT), or aspartate aminotransferase (AST), or alkaline phosphatase (ALP) ≥2X upper limit of normal (ULN), total bilirubin ≥1.5X ULN, or gamma-glutamyl transferase (GGT) ≥3X ULN as per the central laboratory.
20. Estimated glomerular filtration rate (eGFR) at ≤45 mL/min and/or history of persistent micro or macro albuminuria.
21. History of current or prior (within 1 year of Randomization) any significant illness, or any medical history
22. History of bariatric surgery or other surgical or medical history
23. History of current or prior (within 1 year of Randomization) abnormal, clinically significant ECG including inadequately controlled hypertension
24. History or evidence of inherited bleeding diathesis or significant coagulopathy at risk of bleeding.
25. Surgical procedure (including open biopsy, surgical resection, wound revision, or any other major surgery involving entry into a body cavity) or significant traumatic injury
26. Known history of human immune-deficiency virus (HIV), hepatitis C, or hepatitis B infection.
27. Malignancies within 3 years prior to Randomization
28. Donated more than 500 mL of blood or significant blood loss within 60 days before Randomization.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 94 (Actual)
Dates: Start 2023-02-06 (Actual); Primary Completion 2024-04-11 (Actual); Study Completion 2024-04-11 (Actual)

PRIMARY OUTCOMES:
Safety Events | 16 weeks
  Incidence of Adverse Events (AEs) and Serious Adverse Events (SAEs)
Change in Central Subfield Thickness | 12 weeks
  Change from baseline in Central Subfield Thickness (CST), as measured by Spectral Domain Ocular Coherence Tomography (SD-OCT), compared to placebo.

SECONDARY OUTCOMES:
Change in BCVA | 12 weeks
  Change from baseline in Best Corrected Visual Acuity (BCVA) in the Early Treatment Diabetic Retinopathy Study (ETDRS) letter score, compared to placebo.
Change from baseline in Diabetic Retinopathy Severity Score (DRSS), compared to placebo. | 12 weeks
  DRSS is scored on a range from 10 to 90 and where higher scores indicate a worse outcome.
Repeat-dose Cmax of RZ402 | 16 weeks
  Repeat-dose Cmax of RZ402
Repeat-dose T1/2 of RZ402 | 16 weeks
  Repeat-dose T1/2 of RZ402
Repeat-dose AUC of RZ402 | 16 weeks
  Repeat-dose AUC of RZ402

CONTACTS AND LOCATIONS:
Locations (32):
- United States (32):
  - Rezolute Investigative Site, Phoenix, Arizona, Phoenix, Arizona
  - Rezolute Investigative Site, Bakersfield, CA, Bakersfield, California
  - Rezolute Investigative Site, Beverly Hills, California, Beverly Hills, California
  - Rezolute Investigative Site, Fullerton, California, Fullerton, California
  - Rezolute Investigative Site, Modesto, California, Modesto, California
  - Rezolute Investigative Site, Santa Barbara, CA, Santa Barbara, California
  - Rezolute Investigative Site, Coral Springs, Florida, Coral Springs, Florida
  - Rezolute Investigative Site, Deerfield Beach, Florida, Deerfield Beach, Florida
  - Rezolute Investigative Site, Fort Lauderdale, Florida, Fort Lauderdale, Florida
  - Rezolute Investigative Site, Orlando, FL, Orlando, Florida
  - Rezolute Investigative Site, Winter Haven, Florida, Winter Haven, Florida
  - Rezolute Investigative Site, Augusta, Georgia, Augusta, Georgia
  - Rezolute Investigative Site, Oak Forest, Illinois, Oak Forest, Illinois
  - Rezolute Investigative Site, Springfield, IL, Springfield, Illinois
  - Rezolute Investigative Site, Lenexa, KS, Lenexa, Kansas
  - Rezolute Investigative Site, Royal Oak, MI, Royal Oak, Michigan
  - Rezolute Investigative Site, Saint Louis Park, MN, Saint Louis Park, Minnesota
  - Rezolute Investigative Site, Saint Louis, Missouri, St Louis, Missouri
  - Rezolute Investigative Site, Reno, Nevada, Reno, Nevada
  - Rezolute Investigative Site, Bloomfield, NJ, Bloomfield, New Jersey
  - Rezolute Investigative Site, Great Neck, New York, Great Neck, New York
  - Rezolute Investigative Site, New York, New York, New York, New York
  - Rezolute Investigative Site, Springfield, Oregon, Springfield, Oregon
  - Rezolute Investigative Site, Ladson, South Carolina, Ladson, South Carolina
  - Rezolute Investigative Site, Austin, TX, Austin, Texas
  - Rezolute Investigative Site, Bellaire, TX, Bellaire, Texas
  - Rezolute Investigative Site, McAllen, Texas, McAllen, Texas
  - Rezolute Investigative Site, Plano, Texas, Plano, Texas
  - Rezolute Investigative Site, San Antonio, TX, San Antonio, Texas
  - Rezolute Investigative Site, The Woodlands, TX, The Woodlands, Texas
  - Rezolute Investigative Site, Willow Park, Texas, Willow Park, Texas
  - Rezolute Investigative Site, Lynchburg, Virginia, Lynchburg, Virginia

IPD SHARING:
Plan to Share IPD: No